CLINICAL TRIAL: NCT05188625
Title: Comparison of Conventional Face-to-face Dietary Education With Online Self-learning for Women With GDM - a Pilot Study
Brief Title: Online Self-learning for Women With Gestational Diabetes Mellitus
Acronym: iSelf-Learn
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KK Women's and Children's Hospital (Other Government)
Responsible Party: Principal Investigator, Han Wee Meng, Senior Principal Dietitian, Head of Nutrition & Dietetics Department, Principal Investigator, KK Women's and Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019-2927 CIRB
Record Dates: First submitted 2021-11-26; First posted 2022-01-12 (Actual); Last update posted 2022-01-12 (Actual); Status verified 2021-12

CONDITIONS: Gestational Diabetes
Keywords: Gestational Diabetes Mellitus; GDM; Medical Nutrition Therapy; Telehealth
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control arm (No Intervention): This group will receive the standard care of face-to-face dietitian counselling sessions.
- Intervention arm (Experimental): This group will receive online self-paced dietary education, and followed up by telehealth video consultation with dietitian for dietary counselling.
  Interventions: Other: Telesupport - Telehealth

INTERVENTIONS:
Other: Telesupport - Telehealth — Online self-paced dietary education videos; Dietary counselling via video consultation; Blood glucose monitoring via a specially-designed health app
  Arms: Intervention arm

SUMMARY:
This study aims to determine the feasibility and acceptability of using telehealth in the care of women with Gestational Diabetes Mellitus (GDM) by providing a self-learning alternative via an online portal compared to a one-to-one dietary education, conducted face-to-face in a dietitian clinic. The investigators hypothesize that the use of technology would enable a higher percentage of women to receive the necessary dietary education, thereby empowering behaviour change and resulting in positive maternal blood glucose control and pregnancy outcomes.

The primary hypothesis is that the new care model will reach out to a higher proportion compared to the conventional model (Service utilization), as determined by the completion of the online self-learning, comparing it to attendance rates with the conventional model.

The secondary hypothesis is that the new care model will be able to provide care that would be comparable to those in the traditional outpatient clinic setting, as measured by the blood glucose and pregnancy outcomes, as well as patient satisfaction and patient experience.

DETAILED DESCRIPTION:
GDM is a significant health issue amongst women. Medical nutrition therapy is established as the first-line treatment for GDM. The goal is to support maternal and foetal nutrition in order to ensure adequate pregnancy weight gain and foetal growth, whilst at the same time, maintain optimal glycemic control. Health education continues to play an important role in managing GDM. However, not all women with GDM receive dietary education as recommended, due to a multitude of personal and circumstantial factors. Failure to attend diabetes-related appointment has been associated with poorer glycaemic control by 36 weeks' gestation, which leads to a higher risk of macrosomia and an unfavourable set-up for neonatal outcomes. Therefore, this pilot study aims to determine the feasibility and acceptability of using telehealth in the dietary management of GDM compared with the current standard care, i.e. traditional face-to-face dietary education.

A total of 50 women diagnosed with GDM will be randomized to the standard care or telehealth, where self-education will be done via an online portal and subsequently followed up by teleconsult. Both groups will be followed up by the dietitian every 2-4 weeks until delivery either face-to-face (control group) or telehealth video consultation (intervention group). Each participant will be provided with a set of glucometer and the required consumables for home blood glucose monitoring.

Outcomes to determine the success of the study will be the percentage of women who completed dietary education. Other outcomes will include birth outcome data - birth weight to assess for large-for-gestational age baby, type of delivery, incidence of neonatal hypoglycaemia and total maternal weight gain, to establish the efficacy of this model of care. The effectiveness of self-learning will be assessed using pre- and post-test assessment quizzes. The experience and satisfaction of this model will also be surveyed.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy
* Women diagnosed with GDM before 32 weeks
* Women willing and have provided written consent to participate
* Women with ability to use telemedicine services after briefed
* Women who have sufficient communication abilities (written, listening and spoken) to be fully involved
* Women who have access to phone and internet
* Women willing to download and send blood glucose readings to research team.

Exclusion Criteria:

* Multiple pregnancies
* Gestational age 35 weeks and above
* Women with existing Type 1 or Type 2 Diabetes
* Women receiving oral steroid therapy
* Women with evidence of fetal complications (such as fetal anomalies, intrauterine growth retardation) and known history of pregnancy complications (e.g. pre-eclampsia)

Min Age: 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 50 (Actual)
Dates: Start 2021-01-13 (Actual); Primary Completion 2021-06-23 (Actual); Study Completion 2021-08-13 (Actual)

PRIMARY OUTCOMES:
Completion rate | Completion of online dietary education at Day 3
  The completion of online dietary education
Attendance rate | Mean attendance of each dietitian visit throughout study completion for an average of up to 12 weeks.
  The attendance of each dietitian visit

SECONDARY OUTCOMES:
Knowledge assessment using a quiz | At baseline Day 0 and between Day 3 (for intervention group) and Day 14 (for control group)
  The change in knowledge assessment, assessed as difference in score of quiz before and after dietary education
Patient experience | At end of study up to 12 weeks
  The Hospital Consumer Assessment of Healthcare Providers and Systems Survey (HCAHPS) is used to collect information on how satisfied patients are with their healthcare providers; includes questions on level of care & concern, treated with kindness & compassion, courtesy & respect, being listened to
Telehealth usability | At end of study up to 12 weeks
  Usefulness, ease of use, reliability, interface and interaction quality of the telesupport-telehealth service using a specific questionnaire (International Journal of Telerehabilitation 2016; 8(1): 3-10)
Glycaemic control | Every 2-4 weeks throughout the study, up to 12 weeks
  Blood glucose profile ranges pre- and post-meals
Maternal outcome | At end of study, up to 12 weeks
  Total gestational weight gain in kilograms
Foetal outcome 1 | At end of study, up to 12 weeks
  Birth weight in grams
Foetal outcome 2 | At end of study, up to 12 weeks
  Neonatal hypoglycaemia as defined by blood glucose level below 3.0mmol/L

CONTACTS AND LOCATIONS:
Overall Officials: Wee Meng Han, PhD, Principal Investigator — KK Women's and Children's Hospital
Locations (1):
- KK Women's and Children's Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2021-02-10): https://cdn.clinicaltrials.gov/large-docs/25/NCT05188625/Prot_000.pdf
  • Informed Consent Form (2021-02-10): https://cdn.clinicaltrials.gov/large-docs/25/NCT05188625/ICF_001.pdf